CLINICAL TRIAL: NCT06189443
Title: Abdominal-Kegel Exercise in Patients With Stress Urinary Incontinence and the Effect of Telemedicine Applications on Adaptation to Lifestyle Changes: A Randomized Controlled Study
Brief Title: Abdominal-Kegel Exercise and the Effect of Telemedicine in Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Eskisehir City Hospital (Other)
Responsible Party: Principal Investigator, SEVDA SUNGUR, Research Assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EskisehirOU/03.03.2022-20
Record Dates: First submitted 2023-12-09; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; Kegel exercises; Randomization; Telemedicine
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional lifestyle changes and kegel exercise recommended group (No Intervention): Patients with stress urinary incontinence will be given a brochure that will be prepared similar to the brochure given to the Intervention group.
- Group administered to individual telemedicine (Active Comparator): A brochure containing incontinence patient information will be prepared and given, web-based training will be implemented, and informative/reminder messages will be sent via short messages every day.
  Interventions: Other: Group administered to individual telemedicine

INTERVENTIONS:
Other: Group administered to individual telemedicine — A brochure containing incontinence patient information will be prepared and given, web-based training will be implemented, and informative/reminder messages will be sent via short messages every day.
  Other Names: Kegel and abdominal egsercises with telemedicine
  Arms: Group administered to individual telemedicine

SUMMARY:
Urinary incontinence is a very common health problem that reduces the quality of life mostly in women. Behavioral therapy (lifestyle changes, abdominal-Kegel exercises) is recommended as the first choice in the treatment of the disease. It is known that surgical and medical treatment cannot give a definite result. The application of behavioral therapy with telemedicine has advantages such as reducing the cost and increasing the treatment rate. In this study, it is aimed to evaluate the effect of telemedicine practices on compliance with multi-module behavioral therapy in women with stress urinary incontinence.

DETAILED DESCRIPTION:
The study is a randomized controlled study to be conducted in female patients between the ages of 20-65 who applied to the Eskişehir City Hospital urology outpatient clinic and diagnosed with stress urinary incontinence.

When type 1 (α) error was 5%, type 2 error (1-β) was 95%, and the effect size was accepted as 0.5, it was calculated that there should be at least 47 people in the groups.

Stratified and block randomization will be used to recruit patients into study groups.

The patients will be evaluated with the QUID test, risk assessment questionnaire in patients with stress urinary incontinence, incontinence short test, bladder diary, daily urinary incontinence, a notebook to record the duration of the exercises to be performed, quality of life scale and lifestyle changes questioning form.

The intervention group will be re-evaluated as a result of the intervention with measurement tools.

Intervention group: Brochure about incontinence will be given, web-based training will be applied, SMS will be sent every day according to the risks.

Control group: Only brochure will be given.

It is expected that a low-cost application to be developed after the study will reduce the complaints of the patients, increase their quality of life and have a positive effect on women's health.

It is difficult for physicians to allocate sufficient time to convey lifestyle changes and exercises to patients with stress urinary incontinence during their busy work hours in the clinic. After the success to be achieved, the usage rate of the website to be prepared will be increased through various scientific platforms and associations.

ELIGIBILITY:
Inclusion Criteria:

* having symptoms of UI for at least the last 6 months,
* QUID stress score is ≥ 4,
* diagnosed with SUI as a result of the evaluation made by a specialist physician, have minimal skills in using new technologies
* Those who have the opportunity to access the web page to be prepared can participate in the research.

Exclusion Criteria:

* History of using medical therapy for UI,
* existing urinary infection,
* diabetes mellitus,
* nervous system disease (such as multiple sclerosis, cerebrovascular disease),
* psychiatric illness or dementia,
* genitourinary malignancy,
* having limited range of motion in the foot or pelvic region,
* pregnant

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — stress urinary incontinence is common in women than men
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Telemedicine success | 1 year
  Changes in the "frequency of incontinence episodes patients" and "adaptation to lifestyle changes (Body mass index status, smoking, exercise, fluid intake) " in the intervention and control group after the study
Quality of life score | 1 year
  Changes in the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) score. The questionnaire includes questions such as the frequency of urinary incontinence, the amount of leakage, its impact on daily lifestyle, and in what situation the patient leaks urine. The score that can be obtained from the scale is distributed between 0-21. As the total score decreases, the quality of life increases.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Tepebaşı
  - Eskişehir Osmangazi Üniversitesi Tıp Fakültesi, Eskişehir

IPD SHARING:
Plan to Share IPD: No
The information will not be shared as it falls under the personal data protection law.

REFERENCES:
- [Background] Schroeder M, Plotner EA, Sharma S, Hunter K, Spector S, Lipetskaia L. A Randomized Controlled Trial of a Multimedia Patient Education Tool for Stress Versus Urgency Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2021 Jul 1;27(7):403-408. doi: 10.1097/SPV.0000000000000946. PMID 32925421
- [Background] Rygh P, Asklund I, Samuelsson E. Real-world effectiveness of app-based treatment for urinary incontinence: a cohort study. BMJ Open. 2021 Jan 4;11(1):e040819. doi: 10.1136/bmjopen-2020-040819. PMID 33397664